CLINICAL TRIAL: NCT04289545
Title: Postprandial Effects of Functional Bread
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bergen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 11367/2019
Record Dates: First submitted 2020-02-26; First posted 2020-02-28 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-07

CONDITIONS: Postprandial Hyperglycemia
MeSH Terms: conditions — Hyperglycemia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Control Bread (Placebo Comparator): no added guar gum
  Interventions: Dietary Supplement: Functional bread
- Functional Bread 1 (Active Comparator): 10% guar gum, low molecular weight
  Interventions: Dietary Supplement: Functional bread
- functional Bread 2 (Active Comparator): 10% guar gum, high molecular weight
  Interventions: Dietary Supplement: Functional bread
- Functional Bread 3 (Active Comparator): 15% guar gum, low molecular weight
  Interventions: Dietary Supplement: Functional bread
- Functional Bread 4 (Active Comparator): 15% guar gum, high molecular weight
  Interventions: Dietary Supplement: Functional bread

INTERVENTIONS:
Dietary Supplement: Functional bread — Postprandial effects of bread containing galactomannan

SUMMARY:
This study investigates whether bread with added galactomannan, a soluble fiber, can reduce the postprandial glucose response in healthy overweight adults.

DETAILED DESCRIPTION:
This single-blind crossover-designed study wants to investigate the postprandial effect of functional bread in healthy overweight adults. Therefore, four types of bread, consumed by the participants, have added galactomannan in different amounts and viscosities, and one bread is the control bread.

The participants arrive after an overnight fast and before the consumption of bread, a fasting blood sample is taken.

After the ingestion, blood samples are taken at specific times. The area under the curve of the postprandial glucose is expected to differ between the functional breads.

ELIGIBILITY:
Inclusion Criteria:

* healthy, overweight adults (BMI between 25 and 30 kg/m2)

Exclusion Criteria:

* Known diagnosis of diabetes mellitus type 2
* HbA1c at screening ≥ 48 mmol/mol
* Other chronic diseases (heart disease, cancer) within the last 3 years
* Pregnancy and lactation
* Known drug or alcohol abuse
* Unwilling to follow the study requirements

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-07-07 (Actual); Study Completion 2021-07-07 (Actual)

PRIMARY OUTCOMES:
area under the curve of postprandial glucose | 180 minutes

SECONDARY OUTCOMES:
area under the curve postprandial insulin | 180 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Jutta Dierkes, PhD, Principal Investigator — University of Bergen
Locations (1):
- University of Bergen, Research Unit for Health Surveys, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No